CLINICAL TRIAL: NCT04376749
Title: Influence of Caffeine Therapy in Preterm Infants on Sleep and Neurodevelopmental Outcomes During the First Year of Life: a Single Center Experience
Brief Title: Influence of Caffeine Therapy in Preterm Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.950
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Caffeine; Sleep Disorder
Keywords: caffeine,; sleep wake disorder; preterm; neurodevelopment; actigraphy
MeSH Terms: conditions — Sleep Wake Disorders; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preterm infants received caffeine: preterm infants aged between 28 to 34 weeks gestational age who received caffeine therapy either for prophylaxis or treatment
- preterm infants received no caffeine: preterm infants aged between 28 to 34 weeks gestational age who received no caffeine therapy

SUMMARY:
The development of sleep wake cycles is indicative of child's neurocognitive functions. Caffeine therapy is commonly used in neonatal intensive care units for treatment of apnea of prematurity (AOP), to reduce mechanical ventilation, and improve the success of extubation. In addition, it is suggested to be associated with positive long-term outcomes on pulmonary function and neurodevelopment. However, it is still not clear how caffeine therapy affects the sleep architecture and neurodevelopment of preterm infants. Furthermore, optimal dosing and timing of caffeine therapy is controversial.

We aimed to evaluate the effects of caffeine therapy on sleep architecture and neurodevelopment in preterm infants during the first year of life.

A prospective observational case-control study will be conducted. Forty preterm infants aged between 28 to 34 gestational weeks admitted to the Marmara University Neonatal Intensive Care Unit (NICU) from May 2020 to May 2021 will be included. Infants with neonatal risk factors for poor neurodevelopmental outcomes will be excluded. Duration, timing and cumulative dosage of caffeine therapy will be calculated. Follow up outcome for neurodevelopment and sleep architecture of preterm infants who received caffeine therapy will be compared with those who did not receive caffeine therapy.

Sleep and activity behavior recorded by actigraphy, sleep diary and polysomnography at 6, and 12 months corrected age will be compared to noncaffeine group. Neurodevelopment will be assessed by neurological examination defined by Hammersmith, Ages and Stages Questionnaire (ASQ-2), and Bayley Scales of Infant and Toddler Development.

DETAILED DESCRIPTION:
Methylxanthines have been prescribed in preterm infants to treat and prevent Apnea of Prematurity (AOP), for extubation success, for reduction of incidence of BPD, need for treatment of PDA, retinopathy of prematurity, IVH, and for neuroprotective effects. Caffeine is the most common drug of choice. Despite its frequent use there are no standardized protocols for optimal timing and dosage. It is suggested to have a neuroprotective effect, and associated with reduction of neurological disabilities, cognitive delay. However, there are studies which found no difference in poor neurological outcomes compared to control.

Premature infants have more active sleep compared to term infants, and their sleep patterns mature gradually. Studies about the effects of caffeine therapy on sleep of premature infants are few. It is known that sleep is associated with child's neurodevelopmental outcomes. Identifying the impact of caffeine therapy on sleep will help clinicians to identify and improve neurodevelopmental problems in this vulnerable study population.

The aim of this study is to evaluate the effects of caffeine therapy on sleep, activity patterns and neurodevelopment in preterm infants during the first year of life.

Based on the assumption that each year approximately 20 infants receive neonatal caffeine therapy in the unit, forty preterm infants aged between 28 to 34 gestational weeks admitted to the Marmara University Neonatal Intensive Care Unit (NICU) from May 2020 to May 2021 will be included. Duration, timing and cumulative dosage of caffeine therapy will be calculated. The routine practice of Marmara University NICU protocol is to administer caffeine prophylaxis to infants born at less than 30 weeks of gestational age and/or infants with less than 1250 grams gestational weight. Infants born between 30 to 34 weeks of gestational age who has AOP are treated with caffeine therapy with the commonly prescribed dose of 20 mg/kg loading, and 5-10 mg/kg/day maintenance. Neonatal caffeine therapy continues until the infants are 34 weeks corrected gestational age and free of any apnea episodes for at least 7 days. Infants with neonatal risk factors for poor neurodevelopmental outcomes such as infants with perinatal asphyxia, intraventricular hemorrhage grade 3 or higher, retinopathy of prematurity(ROP) of stage 3 or higher, infants using sedative or anticonvulsant drugs at the time of data collection will be excluded.

Follow up outcome for sleep architecture and neurodevelopment of preterm infants who received caffeine therapy will be compared with those who did not receive caffeine therapy.

Actigraphy Sleep and activity behavior recorded by sleep diary, actigraphy and polysomnography at 6, and 12 months corrected age will be compared to noncaffeine group. Sleep wake patterns will be assessed by Philips Respironics Mini-Mitter Actiwatch-2 for at least 3 days at home environment and sleep diaries within 5-minute intervals will be filled out by parents simultaneously. Actigraphy is a validated wristwatch-like device that distinguishes sleep from wakefulness based on accelerometer measured movement. The actiwatch weighs 16 grams and will be placed on the infant's left ankle. For actigraphy interpretation, if the activity count exceeds a predefined threshold value the epoch is scored as wake state. 10 minutes with no movements on autograph will be determined as sleep phase. High frequency movements with >40 movements in each epoch lasting >10 minutes will be determined as wake state. According to the frequency of infants' movements, a number of sleep-wake variables will be calculated for analyses with Philips Actiware 6.1.8 software. Mean total sleep duration, mean sleep duration during the day, mean sleep duration at night, sleep onset latency (SOL: time taken to fall asleep after reported lights out), wake after sleep onset (WASO: number of minutes recorded as wake between sleep onset and sleep offset), longest consolidated sleep period at night (midnight and 6 am), number of night waking, and sleep efficiency (TST/ time in bed, reported as percent) will be determined.

Polysomnography Infants will undergo 3-4 hours polysomnography (Embla Systems N7000) in the pediatric sleep laboratory. Further validation of the actigraphy will be performed by an epoch-by-epoch comparison of actigraphy and simultaneous polysomnography data. The following variables will be monitored: electroencephalography, electromyography, electrocardiography, heart rate and respiratory rate. Respiration will be monitored with a nasal-cannula- pressure transducer, thoracic and abdominal inductive plethysmography bands and pulse-oximetry. Polysomnography will be recorded with Embla RemLogic software. For polysomnography scoring, recommendations of the American Academy of Sleep Medicine Guidelines-2017 will be followed. The polysomnography data will be analyzed by an expert physician blinded to the actigraphy results or the newborn infant's clinical data, except for gestational age and days of life. Apnea-hypopnea index (AHI) will be determined.

Our secondary objective is to assess neurodevelopment of these infants. Neurodevelopment will be assessed by neurological examination defined by Hammersmith, Ages and Stages Questionnaire (ASQ), and Bayley Scales of Infant and Toddler Development at 6, and 12 months corrected age and will be compared to noncaffeine group.

Neurological examination will be performed with Hammersmith Neurological Examination. Hammersmith Neurological Examination is a quick examination for 3 to 24 months old infants. It consists of 26 items assessing neurological function in 5 groups: cranial nerve function (max 15 points), posture (maximum 18 points), movements (maximum 6 points), tone (maximum 24 points) and reflexes and reactions (maximum 15 points). Each subgroup is scored from 0 to 3 points and all scores are summed at the end of the examination.

Ages and Stages Questionnaire helps to evaluate developmental progress in children between the ages of 1 month and 66 months. Ages and Stages Questionnaire lasts approximately 10-15 minutes and assess the child development in 5 developmental areas: gross motor, fine motor, communication, problem solving and personal- social. Each area consists of 6 questions and the questions are answered in 3 simple responses: yes, sometimes or not yet. The questionnaire is scored with a simple 0, 5- and 10-point scoring system (yes: 10 points, sometimes: 5 points, not yet: 0 points) in 2-3 minutes by parents and the results are interpreted according to standardized cutoffs by professionals. Ages and Stages Questionnaire-2 (ASQ-2) is a parent-friendly developmental scale with 0.86 sensitivity, 0.85 specifity, 0.92 test-retest reliability and 0.93 inter-rater reliability. If the score on any domain is <2SDs below the cut-off point for the Turkish reference group, the child is defined as at risk for neurodevelopmental delay.

The Bayley Scales of Infant and Toddler Development, 3rd Edition produces three composite scores: the Cognitive Scale (range 55-145), the Language scale (range 45-155) which has receptive and expressive communication subtests, and the Motor scale (range 45-155), which consists of Fine Motor, and Gross Motor subtests.

Child's scores will be compared to the standardized age norms.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born between 28 to 34 gestational weeks admitted to the Marmara University Neonatal Intensive Care Unit (NICU)

Exclusion Criteria:

* perinatal asphyxia intraventricular hemorrhage grade 3 or higher retinopathy of prematurity(ROP) of stage 3 or higher major congenital anomalies infants using sedative or anticonvulsant drugs at the time of data collection

Ages: 28 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born between 28 to 34 gestational weeks admitted to the Marmara University Neonatal Intensive Care Unit (NICU) during one year period
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Sleep and activity behavior | 6 months corrected age
  Sleep and activity behavior recorded by actigraphy
Sleep and activity behavior | 12 months corrected age
  Sleep and activity behavior recorded by actigraphy
Obstructive Apnea and Hypopnea Index | 6 months corrected age
  Obstrcutive Apnea and Hypopnea Index recorded by Polysomnography
Obstructive Apnea and Hypopnea Index | 12 months corrected age
  Obstrcutive Apnea and Hypopnea Index recorded by Polysomnography

SECONDARY OUTCOMES:
Neurodevelopment | 6 and 12 months corrected age
  Neurological examination by Hammersmith
Neurodevelopment | 6 and 12 months corrected age
  Neurodevelopment assessed by Ages and Stages Questionnaire (ASQ-2)
Neurodevelopment | 6 and 12 months corrected age
  Neurodevelopment assessed by Bayley Scales of Infant and Toddler Development, 3rd edition

CONTACTS AND LOCATIONS:
Overall Officials: Perran Boran, MD, PhD, Principal Investigator — Marmara University
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Atalah YEY, Baris HE, Akdere SK, Sabanci M, Ozdemir H, Gucuyener K, Eralp EE, Ozek E, Boran P. Effects of caffeine therapy for apnea of prematurity on sleep and neurodevelopment of preterm infants at 6 months of corrected age. J Clin Sleep Med. 2023 Dec 1;19(12):2075-2085. doi: 10.5664/jcsm.10760. PMID 37559530